CLINICAL TRIAL: NCT04858906
Title: Neutral Position Facilitates Orotracheal Intubation With Videolaryngoscopes: A Comparing Angulated (McGrath) and Hyperangulated (C-MAC With D-blade) Videolaryngoscopes
Brief Title: Neutral Position Facilitates Orotracheal Intubation With Videolaryngoscopes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to financial issues
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, Principal Investigator,Attending physician of anesthesiology, Mackay Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20MMHIS438e
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Orotracheal Intubation
Keywords: orotracheal intubation; neutral position; sniffing position; video-assisted laryngoscopes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- from neutral to sniffing position (Active Comparator): The patients in this group will be assessed firstly in the neutral position then subsequently in the sniffing position.
  Interventions: Device: McGrath laryngoscope; Device: C-MAC D-blade laryngoscope
- from sniffing position to neutral position (Active Comparator): The patients in this group will be assessed firstly in the sniffing position then subsequently in the neutral position.
  Interventions: Device: McGrath laryngoscope; Device: C-MAC D-blade laryngoscope

INTERVENTIONS:
Device: McGrath laryngoscope — The patients in this group will be evaluated and intubated with McGrath laryngoscope (angulated videolaryngoscope).
Device: C-MAC D-blade laryngoscope — The patients in this group will be evaluated and intubated with C-MAC D-blade laryngoscope (hyperangulated videolaryngoscope).

SUMMARY:
With the advent and more widespread use of video-assisted laryngoscopy (VL), the incidence of difficult intubation has decreased. However, the optimal position for endotracheal intubation facilitated by VL is not yet determined. The objective of this study is to evaluate the effects of different patient positioning (neutral position versus sniffing position) on the glottic view and intubation time during orotracheal intubation facilitated by two video-assisted laryngoscopes (McGrath laryngoscope and C-MAC D-blade laryngoscope). A total of 252 patients who required orotracheal intubation for elective surgery were included in the study. Primary outcomes include airway difficulty score(ADS), intubation difficulty scale (IDS), the percentage of glottic opening (POGO) and intubation time. By the indexes above and crossover analysis, the study aimed to prove the ideal position for VL.

DETAILED DESCRIPTION:
Endotracheal tube general anesthesia (ETGA) is required for a variety of surgeries. Traditionally, the patient is placed in a sniffing position to facilitate endotracheal intubation with a direct laryngoscope. Increased attempts in intubation or intubation failed may be encountered during direct laryngoscope, leading to hypoxemia or neurological sequelae. Injure to the teeth, gingiva or lips is also sometimes unavoidable. With the advent and more widespread use of video-assisted laryngoscopy (VL), the incidence of difficult intubation has decreased.

However, the optimal position for endotracheal intubation facilitated by VL is not yet determined. A previous study suggested that better glottic view is achieved when placing the patient in a neutral position than the sniffing position during orotracheal intubation by fiberoptic bronchoscopy. The objective of this study is to evaluate the effects of different patient positioning (neutral position versus sniffing position) on the glottic view and intubation time during orotracheal intubation facilitated by two video-assisted laryngoscopes (McGrath laryngoscope and C-MAC D-blade laryngoscope).

A total of 252 American Society of Anesthesiologists I-II patients, in the age above 20 years, who required orotracheal intubation for elective surgery were included in the study. Patients received nasotracheal intubation, awake tracheal intubation, emergency surgery, required rapid-sequence intubation (RSI), those in pregnancy, with possible difficult intubation(with oropharyngeal pathology, limited neck mobility, previous head and neck surgical history), anticipated difficult intubation assessed by preoperative Airway Difficult Score(ADS)(≥ 7), with allergy history of common anesthetics agents or any underlying comorbidities which refrain them from receiving common anesthetic agents were excluded.

The types of VL and the orders of position were randomly allocated by computer and the study take place in the operation room. Primary outcomes include airway difficulty (evaluated by ADS), ease of intubation (evaluated by intubation difficulty scale [IDS], the percentage of glottic opening [POGO]) and intubation time. By the indexes above and crossover analysis, the study aimed to prove the ideal position for VL, improve the efficiency of intubation and decrease the rate of difficult intubation by VL in the future.

ELIGIBILITY:
Inclusion Criteria:

* age above 20 years
* Anesthesiologists I-II
* who required orotracheal intubation for elective surgery

Exclusion Criteria:

* nasotracheal intubation
* awake tracheal intubation
* emergency surgery
* required rapid-sequence intubation (RSI)
* those in pregnancy
* with possible difficult intubation(with oropharyngeal pathology, limited neck mobility, previous head and neck surgical history)
* anticipated difficult intubation assessed by preoperative Airway Difficult Score (≥ 7)
* with allergy history of common anesthetics agents
* any underlying comorbidities which refrain them from receiving common anesthetic agents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
airway difficult score (ADS) | Airway difficult score (ADS) is assessed before induction and it take about 3 minutes.
  Airway difficult score (ADS) represents the airway difficulty and it includes thyro-mental distance, Mallampati score, mouth opening, neck mobility and upper incisions. Each element will be scored from 1 to 3 points accordingly. The higher the scores are, the more difficult the airway could be. The minimum value and the maximum value of the airway difficult score (ADS) are 5 and 15 respectively. The definition of possible difficult airway is when the airway difficult score (ADS) score is more than 7 points.
intubation difficulty scale (IDS) | intubation difficulty scale (IDS) is assessed during intubation and the time it take depend on the difficulty of the case.
  Intubation difficulty scale (IDS) represents ease of intubation and it includes times of intubation attempts, numbers of operators, grade of Modified Cormack-Lehane classification, lifting force, laryngeal pressure and vocal cord mobility. Intubation attempts, operators and grade of Modified Cormack-Lehane classification more than one will be scored directly to the numbers accordingly. The other elements will be scored from 0 to 1 point. The higher the scores are, the more difficult the intubation could be. The minimum value of the IDS is 0 and there is no limit of the maximum value. The definition of difficult intubation is when the intubation difficulty scale (IDS) score is more than 6 points.
percentage of glottic opening (POGO) | Percentage of glottic opening (POGO) is evaluated by another anesthesiologist up to 24 hours after intubation ,and it take about 1 minutes.
  Both the glottic views in first position and in second position are evaluated as percentage of glottic opening (POGO) score, ranging from 0 to 100%. The glottic views will be recorded as digital image and be evaluated by another anesthesiologist subsequently.
intubation time | Intubation time is assessed during intubation and the time it take depend on the difficulty of the case.
  Time from when the patient's mouth is opened to the time when intubation is completed and the EtCO2 is detected by the monitor will be recorded.

SECONDARY OUTCOMES:
complications | Tissue injury, sore throat and hoarseness are evaluated in the postoperative period (the day after the surgery). Desaturation or not is assessed during the procedure.
  Complications include tissue injury (injury to the teeth, gingiva or lips), sore throat, hoarseness and desaturation (SpO2<95%), which are recorded as "happened" or "not happened".

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, Bachelor, Principal Investigator — Mackay Memorial Hospital

REFERENCES:
- [Background] Greenland KB, Edwards MJ, Hutton NJ, Challis VJ, Irwin MG, Sleigh JW. Changes in airway configuration with different head and neck positions using magnetic resonance imaging of normal airways: a new concept with possible clinical applications. Br J Anaesth. 2010 Nov;105(5):683-90. doi: 10.1093/bja/aeq239. Epub 2010 Sep 15. PMID 20846964
- [Background] Park S, Lee HG, Choi JI, Lee S, Jang EA, Bae HB, Rhee J, Yang HC, Jeong S. Comparison of vocal cord view between neutral and sniffing position during orotracheal intubation using fiberoptic bronchoscope: a prospective, randomized cross over study. BMC Anesthesiol. 2019 Jan 5;19(1):3. doi: 10.1186/s12871-018-0671-9. PMID 30611215
- [Background] Kang R, Jeong JS, Ko JS, Ahn J, Gwak MS, Choi SJ, Hwang JY, Hahm TS. Neutral Position Facilitates Nasotracheal Intubation with a GlideScope Video Laryngoscope: A Randomized Controlled Trial. J Clin Med. 2020 Mar 2;9(3):671. doi: 10.3390/jcm9030671. PMID 32131521